CLINICAL TRIAL: NCT00232206
Title: A Phase II Study of Cisplatin Plus Docetaxel as Neoadjuvant Therapy for Stages IB Through Selected IIIA NSCLC
Brief Title: Trial of Neoadjuvant Docetaxel and Cisplatin for Resectable Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated due to slow accrual
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other); Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPMC-EACRI-IRB-05-032; IIT #12207
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Non-small-Cell Lung Carcinoma
Keywords: NSCLC; Lung; Cancer; Metastatic; Neoadjuvant; Stage IB Non-Small Cell Lung Cancer (NSCLC); IIA Non-Small Cell Lung Cancer (NSCLC); IIB Non-Small Cell Lung Cancer (NSCLC); Some IIIA Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — Neoadjuvant Therapy; Cisplatin; Docetaxel

INTERVENTIONS:
Drug: Neoadjuvant Therapy with Cisplatin Plus Docetaxel

SUMMARY:
The primary objective of this study is to assess the response rate of treatment with two cycles of cisplatin and docetaxel chemotherapy prior to surgery (neoadjuvant) for early stage non-small cell lung cancer (NSCLC). Secondary objectives of this study include assessment of radiographic response rate by computed tomography (CT) scanning, overall survival, time to progression, rate of complete surgical removal, and adverse reactions. In addition, this study will test whether positron emission tomography (PET) imaging can predict a tumor response. Patients who have a response to chemotherapy may receive 2 additional cycles after recovering from surgery.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for 80% of new lung cancer diagnoses in the US. Surgery is the primary most successful treatment for early stage patients. However, even lung cancers caught at an early stage (stage IB through selected IIIA) have 5 year survivals after surgery at a rate of only 10-60%. Postoperative platinum based chemotherapy offers a 4-15% survival benefit, depending on stage in fit patients after complete surgical removal of early stage disease. Preoperative platinum based chemotherapy has been shown in small randomized trials to benefit patients with stage IIIA, N2 positive disease, but is not standard of care in earlier stage disease, such as the population in this study.

The combination of cisplatin and docetaxel is approved in the US for front line therapy of stage IV NSCLC based on randomized clinical data showing efficacy and manageable toxicity. Given the efficacy and tolerance of this combination in the metastatic setting, this regimen is an obvious choice for study in the neoadjuvant setting.

PET imaging is approved in the US for determining size, site and spread of lung cancer (staging) and has been shown to reduce unnecessary surgery when used as part of preoperative evaluation. Because NSCLC is not 100% responsive to chemotherapy and CT scans may not show a change in tumor size until after several cycles of chemotherapy, PET imaging might be an effective way to provide an earlier and more reliable estimate of response.

Preoperative chemotherapy will be given for a total of two cycles 21 days apart if any adverse events have resolved and there is no evidence of disease progression. Patients will undergo CT chest through liver and PET scans for restaging following the second cycle and will then be scheduled for surgery 3-6 weeks after the second cycle of chemotherapy. Patients who have responded according to CT and/or PET imaging, or surgical pathology will go on to receive an additional two cycles of chemotherapy with docetaxel and cisplatin once the patient has recovered from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC appropriate for surgery
* Medically fit for resection by lobectomy or pneumonectomy
* T1-2N1 disease by CT must have negative N2/N3 nodes by PET
* T3N1 disease must have pathologically negative N2/N3 nodes
* Measurable disease
* Patients must not be receiving other investigational therapy
* Prior surgery for NSCLC okay if resected > or = 5 years prior
* No prior chemotherapy or radiation for NSCLC
* No uncontrolled medical problems
* No factors that would preclude obtaining informed consent
* Age 18 or greater
* Performance status (PS) 0-1
* Peripheral neuropathy must be < grade 1
* Acceptable hematologic and chemistry parameters
* Renal: creatinine clearance (calculated) > 50 cc/min

Exclusion Criteria:

* History of severe hypersensitivity to docetaxel or like drugs
* Pregnant or nursing women
* Prior chemotherapy or radiation for NSCLC
* Symptomatic superior sulcus tumors
* Prior malignancy except for treated non-melanoma skin cancer, in situ cervical cancer, localized prostate cancer or cancer from which the patient has been disease free for greater than three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-11

PRIMARY OUTCOMES:
Primary objective: To assess the pathologic complete and partial response rate to neoadjuvant treatment with two cycles of cisplatin and docetaxel chemotherapy prior to resection of early stage NSCLC

SECONDARY OUTCOMES:
Secondary objectives: Assessment of radiographic response rate by CT scanning, overall survival, time to progression, rate of complete surgical resection and toxicity
Evaluation of the predictive power of PET to define pathologic response

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Director, Lung Research
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States